CLINICAL TRIAL: NCT02122003
Title: Activity and Safety of Second Line SOrafenib After Pazopanib in Patients With Metastatic Renal Cell Carcinoma (SOAP Study)
Brief Title: Second Line Sorafenib After Pazopanib in Patients With RCC
Acronym: SOAP
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: availability of new and more promising therapeutic agents than expected in the experimentation in question
Sponsor: Fondazione IRCCS Istituto Nazionale dei Tumori, Milano (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GP2; Istituto Tumori Milano (Other: Ethical board)
Record Dates: First submitted 2014-04-06; First posted 2014-04-24 (Estimated); Last update posted 2017-11-22 (Actual); Status verified 2017-11

CONDITIONS: Metastatic Renal Cell Carcinoma
Keywords: sorafenib; pazopanib; cross-resistance; TKI; mRCC
MeSH Terms: conditions — Carcinoma, Renal Cell | interventions — Sorafenib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- sorafenib (Experimental): Sorafenib 400 mg bid
  Interventions: Drug: Sorafenib

INTERVENTIONS:
Drug: Sorafenib — Sorafenib 400 mg bid
  Other Names: Nexavar

SUMMARY:
* Retrospective studies showed Sorafenib's efficacy as second line treatment after a Tyrosine Kinase Inhibitor (TKI).
* Currently there is no standard of treatment in 2nd line for patients treated in first line with pazopanib for metastatic Renal Cell Carcinoma (mRCC).
* With this trial we evaluate the efficacy of sorafenib as second line of treatment in patients treated with pazopanib for mRCC.

DETAILED DESCRIPTION:
* Retrospective studies showed Sorafenib's efficacy as second line treatment after a TKI: AXIS study showed sorafenib activity, in terms of Overall Response Rate (ORR), and the absence statistically significant difference in Overall Survival (OS) between the 2 arms, although there is a significant OS increase of 1.4 months in the Axitinib arm. The INTORSECT study (temsirolimus vs sorafenib in 2nd line after sunitinib) didn't demonstrate statistically significant difference for Progression Free Survival (PFS), but it showed an OS increase in patients treated with sorafenib.
* The COMPARZ study demonstrated the non-inferiority of pazopanib vs sunitinib in 1st line of treatment for mRCC.
* Currently there is no standard of treatment in 2nd line for patients treated in first line with pazopanib for mRCC.
* Primary objective:to evaluate the efficacy of sorafenib (PFS) as second line of treatment in patients treated with pazopanib for mRCC.
* Secondary objectives: To evaluate the safety of sorafenib in patients previously treated with pazopanib. To evaluate the Overall Survival. To evaluate the Quality of Life through specific questionnaires (FKSI-19; European Organization for Research and Treatment of Cancer quality of life questionnaire -C30).To assess the predictive role for PFS and OS of arterial blood pressure increase from baseline to week 4 and 8 after start of treatment with sorafenib. To assess the predictive role for PFS and OS of hand-foot syndrome before week 4 and 8 after start of treatment with sorafenib.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Patients with histological diagnosis of Renal Cell Carcinoma (RCC)
* Measurable disease
* Eastern Cooperative Oncology Group (ECOG) Performance Status of 0 or 1
* Life expectancy of at least 12 weeks.
* Adequate bone marrow, liver and renal function as assessed by the following laboratory requirements to be conducted within 7 days prior to screening:

  * Hemoglobin >= 10.0 g/dl
  * Absolute neutrophil count (ANC) >1,500/mm3
  * Platelet count >= 100,000/ml
  * Total bilirubin ≤ 1.5 times the upper limit of normal
  * ALT and AST ≤ 2.5 x upper limit of normal
  * Alkaline phosphatase ≤ 4 x upper limit of normal
  * prothrombin time-international normalized ratio /partial thromboplastin time ≤ 1.5 x upper limit of normal [Patients who are being therapeutically anticoagulated with an agent such as coumadin or heparin will be allowed to participate provided that no prior evidence of underlying abnormality in these parameters exists.] For patients on warfarin, close monitoring of at least weekly evaluations will be performed, until international normalized ratio is stable based on a measurement at pre-dose, as defined by the local standard of care.
* Prognosis according to Heng: good or intermediate
* Previous treatment with pazopanib
* Pregnant or breast-feeding patients. Women of childbearing potential must have a negative pregnancy test performed within 7 days of the start of treatment. Both men and women enrolled in this trial must use adequate barrier birth control measures during the course of the trial and two weeks after the completion of trial.
* Signed informed consent must be obtained prior to any study specific procedures

Exclusion Criteria:

* First line treatment for metastatic RCC other than pazopanib.
* History of cardiac disease: congestive heart failure >New York Heart Association class 2; active CAD (MI more than 6 mo prior to study entry is allowed); cardiac arrhythmias requiring anti-arrhythmic therapy (beta blockers or digoxin are permitted) or uncontrolled hypertension (>= 160 mmHg systolic and/or 90 mmHg diastolic).
* History of HIV infection
* Active clinically serious infections (> grade 2 NCI-CTC version 3.0)
* Brain or meningeal metastases
* Patients with seizure disorder requiring medication (such as steroids or anti-epileptics)
* History of organ allograft
* Patients with evidence or history of bleeding diathesis
* Patients undergoing renal dialysis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2016-09; Primary Completion 2017-11-08 (Actual); Study Completion 2017-11-08 (Actual)

PRIMARY OUTCOMES:
Progression Free Survival (months) of patients treated with sorafenib after progression to pazopanib | 24 months

SECONDARY OUTCOMES:
Safety profile of sorafenib using Common Terminology Criteria for Adverse Events (CTCAE) criteria v.4.0 in patients previously treated with pazopanib | 24 months
Overall Survival (months) of patients treated with sorafenib after pazopanib progression | 24 months
Quality of Life of patients treated with sorafenib after pazopanib progression using the specific questionnaires FKSI-19 and European Organization for Research and Treatment of Cancer quality of life questionnaire -C30. | 24 months

CONTACTS AND LOCATIONS:
Locations (1):
- Istituto Tumori, Milan, Mi, Italy

REFERENCES:
- [Derived] Iacovelli R, Verzoni E, Grassi P, Farcomeni A, de Braud F, Procopio G. Rationale and protocol of SOAP: a phase II study to evaluate the efficacy of sorafenib as second-line treatment after pazopanib in patients with advanced renal cell carcinoma. Tumori. 2014 Nov-Dec;100(6):e282-5. doi: 10.1700/1778.19296. PMID 25688511